CLINICAL TRIAL: NCT05349708
Title: Benefit of a Telehealth Home-monitoring Program for Vulnerable Patients and Patients Living With Frailty Undergoing Heart Surgery
Brief Title: Telehealth Home-monitoring for Frailty in Cardiac Surgery
Acronym: THE-FACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Brunswick Heart Centre (Other)
Responsible Party: Principal Investigator, Dr. Jean-François Légaré, Clinical Head of Cardiac Surgery, New Brunswick Heart Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 100097
Record Dates: First submitted 2022-04-06; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Frailty; Surgery; Cardiac Event
Keywords: technology; outcomes; hospital readmission; feasibility; follow-up; remote care
MeSH Terms: conditions — Frailty; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant (Experimental): Patients who were sent home with the intervention post-surgery
  Interventions: Device: THE-FACS
- Historical controls (No Intervention)

INTERVENTIONS:
Device: THE-FACS — Telehealth home-monitoring tablet and blood pressure cuff
  Arms: Participant

SUMMARY:
Cardiac surgical interventions are increasingly offered to vulnerable patients or patients living with frailty. Unfortunately, frailty has been shown to be an independent predictor of poorer outcome and increased health care resources in terms of readmission to hospital or visit to the ER after discharge. We hypothesize that the use of a comprehensive Telehealth home-monitoring program could reduce emergency room visits and re-hospitalization after heart surgery.

Frailty in all patients will be determined using the Edmonton frailty scale (EFS) as is part of the current standard of care for all patients at the NBHC since 2018. We plan to implement the Telehealth intervention on all 120 consecutively enrolled patients identified as vulnerable and/or frail and discharged from hospital within 10 days of their surgery. The primary outcome of interest will be rates of ER visit and readmission to hospital within 30 days of discharge compared to propensity score matched historical control patients. A power calculation suggests that 120 patients per group are necessary explaining why the intervention group will be 120 patients. We chose to compare our intervention to a matched group of 240 individuals from historical data which already captures follows patients 30 days after surgery but is limited in its Telehealth intervention. Duration of the study is 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, aged 55 years or older, undergoing elective isolated coronary artery bypass grafting (CABG), aortic valve repair/replacement, mitral valve repair/replacement or combined CABG/valve procedures.
2. Patients defined as pre- vulnerable, vulnerable or frail based on the Edmonton frailty scale (> 4 considered pre- vulnerable) as defined prior to surgery

Exclusion Criteria:

1. Medical reasons for exclusion

   1. Patients who have unstable or recent unstable cardiac syndrome requiring urgent (within 24hr) or emergent surgery
   2. Acute endocarditis who are at higher risk for adverse events
2. Dialysis dependent who are at higher risk for adverse events
3. Patients who have cognitive deficits, visual impairments, inability to read or major difficulties with electronic devices that would preclude use of the intervention
4. Patients who do not have any support or potential caregivers to help facilitate their transition home
5. Patients undergoing minimally invasive surgery which has been shown to enhance recovery
6. Patients unable to be discharged home within 10 days of their surgery. The average length of hospitalization is 5 days with frail patients often requiring additional time but usually within 10 days unless some major barrier exists in allowing discharge home.
7. Patients who are transferred to another hospital for recovery or care.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Rates of emergency room visit and readmission to hospital | 30 days of discharge post-cardiac surgery
  The aim was to compare the rate of emergency room visits and readmission to hospital within 30 days of discharge between two groups of patients: frail, post-surgery cardiac surgery patients who went home with the intervention for self-monitoring of health versus historical controls

SECONDARY OUTCOMES:
Length of hospital stay (LOS, days) and discharge disposition | Duration of stay at the hospital post-cardiac surgery
  The post-surgery inclusion criterion was the LOS of 10 days or less and home-discharge. The investigators, therefore, assessed the LOS and discharge disposition of the frail participants who consented to participate in the study to understand the challenges in recovery and ability to participate in the study.
Rate of readmission to hospital and/or ER visit and reasons | 30 days of discharge post-cardiac surgery
  The aim of the telehealth home monitoring platform was to reduce hospital readmission and/ or ER visits within 30 days of discharge post-cardiac surgery. The investigators, therefore, wanted to explore the rates and causes for the above-mentioned outcomes.
Percentage of patients who faced difficulties with the Telehealth intervention and causes of the same | 30 days of discharge post-cardiac surgery
  Identification of the major challenges frail participants faced in using a technology-based home monitoring program to self-monitor their health and recovery post-cardiac surgery. A participation-satisfaction questionnaire was used to assess the percentage of patients who could/ count not use the intervention and the reasons for such (technological challenges, connectivity ussies, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Légaré, M.D., Ph.D., Principal Investigator — New Brunswick Heart Centre
Locations (1):
- New Brunswick Heart Centre, Saint John Regional Hospital, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No